CLINICAL TRIAL: NCT05919186
Title: Impact of Repeated Antioxidant Supplementation of Embryo Culture Media on Blastocyst Utilization and Expansion Rate Under Two Different O2 Concentrations
Brief Title: Effects of Antioxidant Supplementation of Culture Media on IVF Embryos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liliana Berenice Ramírez Domínguez (Industry)
Responsible Party: Sponsor-Investigator, Liliana Berenice Ramírez Domínguez, Scientific Coordinator, Center of Innovation Technology & Reproductive Medicine
Organization: Center of Innovation Technology & Reproductive Medicine (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CI-20-102
Record Dates: First submitted 2023-05-12; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Infertility, Female; Infertility, Male
Keywords: Blastocyst Rate; IVF; Embryo Culture; Antioxidants
MeSH Terms: conditions — Infertility, Female; Infertility, Male

STUDY DESIGN:
Intervention Model Description: The data registry utilized internal and external measures to ensure accuracy. SOPs were developed for registry operations and data analysis. Data were recorded in clinical records and clinic-specific databases. Regular backups and monthly audits were conducted to safeguard data and verify accuracy. External audits occurred every 6 months. Access controls protected privacy. Appropriate statistical techniques and sample size assessment were used for data analysis. A study on embryo development analyzed 3603 zygotes, assessing blastocyst outcomes and detailing procedures for ovarian stimulation, retrieval, sperm preparation, and assisted reproduction techniques. These measures ensured accurate and reliable results.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EmrbyORP continued at high O2 (Experimental): Antioxidants supplementation Every 12 hours (3.5 μL)
  Interventions: Drug: EmbryORP®; Device: O2 tension 20%
- EmrbyORP at baseline with high O2 (Experimental): Antioxidants supplementation At baseline only (6.5 μL)
  Interventions: Drug: EmbryORP®; Device: O2 tension 20%
- EmrbyORP continued at low 02 (Experimental): Antioxidants supplementation Every 12 hours (3.5 μL)
  Interventions: Drug: EmbryORP®; Device: O2 tension 5%
- EmrbyORP at baseline with low o2 (Experimental): Antioxidants supplementation At baseline only (6.5 μL)
  Interventions: Drug: EmbryORP®; Device: O2 tension 5%

INTERVENTIONS:
Drug: EmbryORP® — EmbryORP® is a novel antioxidant (Cystein 32.9 mM, Glutation 32.6 mM, Ascorbic Acid 22.7 mM)
  Other Names: EmbryORP
Device: O2 tension 20% — After fertilization check, zygotes were placed in the incubator at 37°C, 8% CO2, and 95%
  Arms: EmrbyORP at baseline with high O2; EmrbyORP continued at high O2
Device: O2 tension 5% — After fertilization check, zygotes were placed in the incubator at 37°C, 8% CO2 and 95%
  Arms: EmrbyORP at baseline with low o2; EmrbyORP continued at low 02

SUMMARY:
The goal of this clinical trial is to investigate the impact of repeated antioxidant supplementation on blastocyst utilization and expansion rates in embryos under different oxygen concentrations. The study aims to answer the following main questions:

* Does adding antioxidants every 12 hours to embryo culture media improve usable and expanded blastocyst utilization rates on days 5 and 6?
* How are the O2 concentrations related to the effect of different methods of antioxidants supplementation on blastocysts utilization and expansion rates?

Participants in this study are infertile couples undergoing in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) cycles.

* Zygotes will be incubated at either 5% or 20% oxygen tension until the blastocyst stage.
* Sibling zygotes will be divided into four groups: Group 1A and 1B: Antioxidants every 12 hours at either 5% or 20% O2 tension, respectively. Group 2A and 2B: Antioxidants only once at the beginning of embryo culture at either 5% or 20% O2 tension, respectively.

Researchers will compare the four groups to determine if the repeated antioxidant supplementation of the culture media leads to improved blastocyst utilization and expansion rates compared to the baseline group.

DETAILED DESCRIPTION:
This study is focused on the role of antioxidants (AOXs) in mitigating reactive oxygen species and oxidative stress, which have been associated with failure in in vitro fertilization (IVF) and intracytoplasmic sperm injection (ICSI). The research aimed to evaluate the effect of two different methods of antioxidants supplementation at two O2 tensions on blastocyst utilization and expansion rates. To achieve this, 3603 zygotes from infertile couples undergoing IVF or ICSI were included in the study. The zygotes were divided into two groups: Group 1A and 1B: Antioxidants every 12 hours at either 5% or 20% O2 tension, respectively. Group 2A and 2B: Antioxidants only once at the beginning of embryo culture at either 5% or 20% O2 tension, respectively.

.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women with from 18 to 37 years old at the moment of oocyte collection, tubal factor, polycystic ovary syndrome, uterine factor, or unexplained infertility.
* More than 2 oocytes by conventional in vitro fertilization (cIVF) and intracytoplasmic sperm injection (ICSI).

Exclusion Criteria:

* Infertile woman in assisted reproduction treatment with less than 2 oocytes collected.
* Infertile woman in assisted reproduction treatment with less than 2 oocytes fertilized by conventional in vitro fertilization (cIVF) and intracytoplasmic sperm injection (ICSI)

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 293 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Rate of usable blastocysts on day 5 | 5 days
  Usable blastocysts were defined as vitrified, transferred, and/or biopsied blastocysts at day 5
Rate of expanded blastocysts on day 5 | 5 days
  Expanded blastocysts were defined as usable blastocysts with a 4 to 6 expansion grade at day 5
Rate of sable blastocysts on day 6 | 6 days
  Usable blastocysts were defined as vitrified, transferred, and/or biopsied blastocysts at day 6
Rate of expanded blastocysts on day 6 | 6 days
  Expanded blastocysts were defined as usable blastocysts with a 4 to 6 expansion grade at day 6
Rate of acumulative usable blastocysts | 5 - 6 days
  Usable blastocysts were defined as vitrified, transferred, and/or biopsied blastocysts at days 5 and 6
Rate of acumulative expanded blastocysts. | 5 - 6 days
  Expanded blastocysts were defined as usable blastocysts with a 4 to 6 expansion grade at days 5 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Agarwal, PhD, Study Director — Global Andrology Forum
Locations (1):
- CITMER, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khalied Kaskar, C. Optimizing embryo culture conditions and spent culture media analysis as predictors of em-bryo quality and pregnancy; PhD Thesis, University of the West Cape, Cape Town, South Africa, February 2021.
- [Background] Swain JE. Optimizing the culture environment in the IVF laboratory: impact of pH and buffer capacity on gamete and embryo quality. Reprod Biomed Online. 2010 Jul;21(1):6-16. doi: 10.1016/j.rbmo.2010.03.012. Epub 2010 Mar 21. PMID 20570214
- [Background] Lane M, Lyons EA, Bavister BD. Cryopreservation reduces the ability of hamster 2-cell embryos to regulate intracellular pH. Hum Reprod. 2000 Feb;15(2):389-94. doi: 10.1093/humrep/15.2.389. PMID 10655311
- [Background] Nastri CO, Nobrega BN, Teixeira DM, Amorim J, Diniz LMM, Barbosa MWP, Giorgi VSI, Pileggi VN, Martins WP. Low versus atmospheric oxygen tension for embryo culture in assisted reproduction: a systematic review and meta-analysis. Fertil Steril. 2016 Jul;106(1):95-104.e17. doi: 10.1016/j.fertnstert.2016.02.037. Epub 2016 Mar 21. PMID 27012651
- [Background] Edwards LJ, Williams DA, Gardner DK. Intracellular pH of the preimplantation mouse embryo: effects of extracellular pH and weak acids. Mol Reprod Dev. 1998 Aug;50(4):434-42. doi: 10.1002/(SICI)1098-2795(199808)50:43.0.CO;2-J. PMID 9669527
- [Background] Hong KH, Lee H, Forman EJ, Upham KM, Scott RT Jr. Examining the temperature of embryo culture in in vitro fertilization: a randomized controlled trial comparing traditional core temperature (37 degrees C) to a more physiologic, cooler temperature (36 degrees C). Fertil Steril. 2014 Sep;102(3):767-73. doi: 10.1016/j.fertnstert.2014.06.009. Epub 2014 Jul 17. PMID 25044079
- [Background] Chui, A.; Kalionis, B.; Brennecke, S.; Murthi, P. 201 Homeobox Gene DLX3 Regulates Forskolin Induced Tropho-blast Differentiation. Reprod Fertil Dev 2008, 20(9), 1-1
- [Background] Agarwal A, Gupta S, Sharma RK. Role of oxidative stress in female reproduction. Reprod Biol Endocrinol. 2005 Jul 14;3:28. doi: 10.1186/1477-7827-3-28. PMID 16018814
- [Background] Carocho M, Ferreira IC. A review on antioxidants, prooxidants and related controversy: natural and synthetic compounds, screening and analysis methodologies and future perspectives. Food Chem Toxicol. 2013 Jan;51:15-25. doi: 10.1016/j.fct.2012.09.021. Epub 2012 Sep 24. PMID 23017782
- [Background] Guerin P, El Mouatassim S, Menezo Y. Oxidative stress and protection against reactive oxygen species in the pre-implantation embryo and its surroundings. Hum Reprod Update. 2001 Mar-Apr;7(2):175-89. doi: 10.1093/humupd/7.2.175. PMID 11284661
- [Background] Budani MC, Tiboni GM. Effects of Supplementation with Natural Antioxidants on Oocytes and Preimplantation Embryos. Antioxidants (Basel). 2020 Jul 12;9(7):612. doi: 10.3390/antiox9070612. PMID 32664650
- [Background] Coria-Gomez CR, Torres-Rodriguez P, Villar-Munoz LG, Jimenez-Medina I, Agarwal A, Henkel R, Maldonado-Rosas I, L Trevino C. Comparative study of fertility parameters in vitrified human spermatozoa in the presence or absence of EmbryORP(R) : A novel antioxidant. Andrologia. 2021 May;53(4):e13886. doi: 10.1111/and.13886. Epub 2021 Feb 7. PMID 33550605
- [Background] David Gardner; William Schoolcraft. In Vitro Culture of Human Blastocysts. In Towards Reproductive Certainity: Fertility and Genetics Beyond 1999: The Plenary Proceedings of the 11th World Congress on In Vitro Fertilization & Hu-man Reproductive Genetics; Jansen, R., Mortimer, D., Eds.; Parthenon Publishing Group: London, 1999; Vol. 1, pp. 378-388.
- [Background] Sallam, N.; Hegab, M.; Mohamed, F.; El-Kaffash, D. Effect of Oxidative Stress in Semen, Follicular Fluid and Em-bryo Culture Medium on the Outcome of Assisted Reproduction. Al-Azhar Internat Med J 2021, 2(7), 59-65, doi:10.21608/aimj.2021.79536.1495
- [Background] Truong T, Gardner DK. Antioxidants improve IVF outcome and subsequent embryo development in the mouse. Hum Reprod. 2017 Dec 1;32(12):2404-2413. doi: 10.1093/humrep/dex330. PMID 29136144
- [Background] Bedaiwy MA, Falcone T, Mohamed MS, Aleem AA, Sharma RK, Worley SE, Thornton J, Agarwal A. Differential growth of human embryos in vitro: role of reactive oxygen species. Fertil Steril. 2004 Sep;82(3):593-600. doi: 10.1016/j.fertnstert.2004.02.121. PMID 15374701
- [Background] Bedaiwy M, Agarwal A, Said TM, Goldberg JM, Sharma RK, Worley S, Falcone T. Role of total antioxidant capacity in the differential growth of human embryos in vitro. Fertil Steril. 2006 Aug;86(2):304-9. doi: 10.1016/j.fertnstert.2006.01.025. Epub 2006 Jun 12. PMID 16769062
- [Background] Gardner DK, Kuramoto T, Tanaka M, Mitzumoto S, Montag M, Yoshida A. Prospective randomized multicentre comparison on sibling oocytes comparing G-Series media system with antioxidants versus standard G-Series media system. Reprod Biomed Online. 2020 May;40(5):637-644. doi: 10.1016/j.rbmo.2020.01.026. Epub 2020 Feb 5. PMID 32299733
- [Background] Majumdar G, Majumdar A, Verma IC, Upadhyaya KC. Relationship Between Morphology, Euploidy and Implantation Potential of Cleavage and Blastocyst Stage Embryos. J Hum Reprod Sci. 2017 Jan-Mar;10(1):49-57. doi: 10.4103/0974-1208.204013. PMID 28479756
- [Background] Swain JE. Media composition: pH and buffers. Methods Mol Biol. 2012;912:161-75. doi: 10.1007/978-1-61779-971-6_10. PMID 22829374
- [Background] Agarwal A, Majzoub A. Role of Antioxidants in Assisted Reproductive Techniques. World J Mens Health. 2017 Aug;35(2):77-93. doi: 10.5534/wjmh.2017.35.2.77. Epub 2017 Apr 30. PMID 28497913

DOCUMENTS (3):
  • Study Protocol (2021-10-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT05919186/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT05919186/SAP_001.pdf
  • Informed Consent Form (2021-10-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT05919186/ICF_002.pdf